CLINICAL TRIAL: NCT02882308
Title: Phase II(Window) Preoperative Study of Olaparib With Cisplatin or With Durvalumab (MEDI4736) or Alone or no Treatment in Patients With Histologically Proven Squamous Cell Carcinoma of the Head and Neck Who Are Candidates for Surgery.
Brief Title: Preoperative Administration of Olaparib With Cisplatin or With Durvalumab or Alone or no Tratment in Patients Who Are Candidates for Surgery of Carcinoma of the Head and Neck.
Acronym: OPHELIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HE5A/15; 2015-005268-41 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-08-29 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — olaparib; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Monotherapy with olaparib (Experimental): Patients in the monotherapy arm will be treated with olaparib until the 21st -28th day depending on the day of surgery, will be reassessed by imaging (tumour objective response by RECIST) on the 22nd -28th day and then have a second biopsy or be operated on the 23rd - 29th day. If surgery is delayed, olaparib will be continued until the day before surgery.
  Interventions: Drug: Olaparib
- Combination of cisplatin and olaparib (Experimental): Patients in the cisplatin - olaparib combination arm will receive treatment until the 5th day, will be reassessed by imaging (tumour objective response by RECIST) on the 22nd -28th day and then will have a second biopsy or be operated on the 23rd - 29th day.
  Interventions: Drug: Olaparib; Drug: Cisplatin
- No treatment arm (No Intervention): Patients in the "no treatment" arm will wait to be operated or have a second biopsy on the 23rd - 29th day.Optionally, patients who have a baseline FDG-PET/CT scan may be re-examined on the 22nd -28th day by the same modality to assess metabolic response.
- Combination of durvalumab and olaparib (Experimental): Patients in the durvalumab - olaparib combination arm will receive treatment until the 21th-28th day, will be reassessed by imaging (tumour objective response by RECIST) on the 22nd -28th day and then will have a second biopsy or be operated on the 23rd - 29th day. If surgery is delayed, olaparib will be continued until the day before surgery.
  Interventions: Drug: Olaparib; Drug: Durvalumab

INTERVENTIONS:
Drug: Olaparib — 50/25 mg BD split x 5 days
  Other Names: Lynparza
  Arms: Combination of cisplatin and olaparib
Drug: Cisplatin — 60 mg/m^2 d1-d5
  Other Names: Platamine
  Arms: Combination of cisplatin and olaparib
Drug: Olaparib — 300 mg BD x 21-28 days.
  Other Names: Lynparza
  Arms: Combination of durvalumab and olaparib; Monotherapy with olaparib
Drug: Durvalumab — 1500 mg d1
  Other Names: Imfinzi
  Arms: Combination of durvalumab and olaparib

SUMMARY:
OPHELIA (OPHELIA (OlaParib and durvalumab in HEad and neck squamous celL carcInomA) trial is a Greek, investigator-initiated, randomized open-label window-of-opportunity phase II study. Patients with operable histologically documented squamous-cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx will be randomized between combination with durvalumab and olaparib, cisplatin and olaparib, monotherapy with olaparib or no treatment, before starting standard treatment.

DETAILED DESCRIPTION:
OPHELIA is a window-of-opportunity phase II study randomized between combination with durvalumab and olaparib, cisplatin and olaparib, monotherapy with olaparib or no treatment, before starting standard treatment.

Although patients will be randomized between the 4 arms, no formal comparison between the 4 arms will be performed.Patients allocated to the olaparib monotherapy arm will serve as a proof-of-concept to interpret the mechanism of action of olaparib. Patients allocated in the "no treatment" group will be used as control.

The primary endpoint will be the change in the tumour Ki-67 before and after treatment with the combination of olaparib + durvalumab or olaparib + cisplatin or olaparib monotherapy. Secondary endpoints will be early tumour response by RECIST criteria, pathologic complete response rate, tolerability to treatment and surgical complications rate, and optionally, metabolic response assessed by FDG-PET/CT scan. Translational correlates will be tested in tumour tissue, plasma and germline DNA.

All the endpoints will be analyzed by an "as treated analysis" since the trial does not include a formal comparison of the treatment arms.

Administration of olaparib monotherapy has been associated with reports of the following laboratory findings and/or clinical diagnoses, generally of mild or moderate severity (CTCAE Grade 1 or 2) and generally not requiring treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent prior to any study specific procedures
2. Female and/or male patients aged 18 years and over
3. Body weight higher than 30 Kg
4. Newly diagnosed histologically proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx
5. Provision of biological material (tumor tissue and blood), provision of signed informed consent for translational research
6. Patients selected for a primary surgical treatment
7. No prior anti-cancer treatment for head and neck cancer
8. Performance status ECOG 0-1
9. Adequate hematological status: neutrophils (ANC) ≥1.5x109/L; platelets ≥100x109/L; haemoglobin ≥10g/dL
10. Adequate renal function: serum creatinine level 1.5 mg/dl and Glomelular Filtration Rate50 ml/min by Cockroft/Gault formula
11. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase, AST (SGOT), ALT (SGPT) 5xULN
12. No active rheumatoid arthritis, active inflammatory bowel disease, chronic infections, or any other disease or condition associated with chronic inflammation.
13. Ability to swallow tablets.
14. Regular follow-up feasible
15. Baseline evaluations performed before registration: clinical and blood evaluations no more than 1 week (7 days) prior to registration, tumour assessment (CT or MRI scan of the head and neck, chest, abdomen and pelvis at the discretion of the investigator) no more than 30 days prior to registration
16. Treatment initiation planned less than 1 week (7 days) after registration
17. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if theyhave been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). For female patients of childbearing potential, negative serum pregnancy test within 1 week (7 days) prior of starting study treatment
18. Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination, throughout the period of taking study treatment and for at least 1-6 month (according to the treatment group) after last dose of study drug(s) (where applicable). Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of TWO highly effective forms of contraception in combination, throughout the period of taking study treatment and for 3- 6 months (according tot he treatment group) after last dose of study drug(s) (where applicable).

Exclusion Criteria:

1. Metastatic or locally advanced unresectable disease
2. Uncontrolled hypercalcemia
3. Concomitant unplanned antitumour therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy)
4. Treatment with any other investigational medicinal product within 28 days prior to study entry
5. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
6. Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IMP and up to 30 days after the last dose of IMP.
7. Treatment with CYP3A4 inhibitors as well as inducers, unless discontinued 7 days prior to randomization
8. Any of the following within 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding, treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis
9. Other concomitant or previous malignancy, except: i) adequately treated in-situ carcinoma of the uterine cervix, ii) basal or squamous cell carcinoma of the skin, iii) cancer in complete remission for 5 years
10. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
11. Pregnant or breastfeeding women
12. Patients with known allergy to any excipients to study drugs
13. History of myocardial infarction and/or stroke or other arterialthrombotic events or pulmonary embolism or unstable angina pectoris within 6 months prior to registration
14. No features suggestive of myelodysplastic syndrome/ acute myeloid leukemia MDS/ AML
15. Poorly controlled cardiac arrhythmias
16. Lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, bowel obstruction or inability to take oral medication
17. Active rheumatoid arthritis, active inflammatory bowel disease, chronic infections, or any other disease or condition associated with chronic inflammation.
18. History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan
19. Other clinically significant disease or co-morbidity which may adversely affect the safe delivery of treatment within this trial
20. Known history of positive tests for human immunodeficiency virus (HIV) infection, hepatitis A or C virus, acute or chronic active hepatitis B infection
21. History of severe tumour bleeding or bleeding disorders
22. No blood transfusion within the 28 days prior to study
23. Poorly controlled anti-coagulation therapy (INR3.0 on coumadin or heparin compounds)
24. Palliative radiation therapy within 4 weeks prior to registration
25. Pregnancy or men or women of reproductive age not agreeing to use contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Investigation of the change in the tumour Ki-67 before and after treatment with the combination of olaparib + durvalumab or olaparib + cisplatin or olaparib monotherapy. | At baseline and at the day of the surgery or 2nd biopsy (at days 23-29 days)

SECONDARY OUTCOMES:
Objective response rate according to RECIST 1.1 criteria | Imaging studies will be performed at baseline and on week 4
Pathologic complete response rate | On week 4 only for operable patients
Metabolic response rate assessed by FDG-PET/CT scan (optional) | At baseline, on week 4
Number of participants with tolerability to the treatment. | From the 1st day of therapy and every week for 4 weeks maximum and 90 days after last therapy administration
Surgical complication rate | Up to 30 days after surgery or the day of initiation of the next anticancer therapy
Mutations in genes associated with DNA repair | At baseline, on day of surgery or the 2nd biopsy (at days 23-29)
Expression of tissue biomarker: PARP1 | At baseline, on day of surgery or the 2nd biopsy (at days 23-29)
Expression of tissue biomarker: BRACA1,2 | At baseline, on day of surgery or the 2nd biopsy (at days 23-29)
Expression of tissue biomarker: ERCC1 | At baseline, on day of surgery or the 2nd biopsy (at days 23-29)
Expression of tissue biomarker: PDL-1 | At baseline, on day of surgery or the 2nd biopsy (at days 23-29)
Expression of tissue biomarker: TILs | At baseline, on day of surgery or the 2nd biopsy (at days 23-29)
Plasma methylation biomarker: PARP1 methylation in plasma cell-free DNA | At baseline, a day before surgery and 90 days after surgery
Plasma methylation biomarker: BRCA1,2 methylation in plasma cell-free DNA | At baseline, a day before surgery and 90 days after surgery
Plasma methylation biomarker: ERCC1 methylation in plasma cell-free DNA | At baseline, a day before surgery and 90 days after surgery
Plasma methylation biomarker: RAD51C methylation in plasma cell-free DNA | At baseline, a day before surgery and 90 days after surgery
Single-nucleotide polymorphisms: PARP-1 Val762Ala | Sample will be collected once at baseline
Single-nucleotide polymorphisms: ERCC1 Asn118Asn (C/T) | Sample will be collected once at baseline
Single-nucleotide polymorphisms:ERCC2 Lys751Gln (T/G) | Sample will be collected once at baseline
Single-nucleotide polymorphisms: GSTP1 Ile105Val (A/G) | Sample will be collected once at baseline
Single-nucleotide polymorphisms: XPD Lys751Gln (A/C, C/C) | Sample will be collected once at baseline
Single-nucleotide polymorphisms: XRCC1 Arg399Gln (G/A) | Sample will be collected once at baseline
Circulating tumor cells (CTCs) evaluated for DNA repair biomarkers | At baseline, a day before surgery and 90 days after surgery
Circulating tumor cells (CTCs) evaluated for PD-L1 | At baseline, a day before surgery and 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diamanto Psyrri, MD,Ass.Prof, Principal Investigator — Division of Oncology, 2nd Dept of Internal Medicine, University Hospital "Attiko"
Locations (2):
- Greece (2):
  - Euromedica General Clinic of Thessaloniki, Thessaloniki, Thessaloniki
  - University Hospital "Attikon", 2nd Department of Internal Medicine, Division of Oncology, Athens

REFERENCES:
- [Derived] Psyrri A, Gkotzamanidou M, Papaxoinis G, Krikoni L, Economopoulou P, Kotsantis I, Anastasiou M, Souliotis VL. The DNA damage response network in the treatment of head and neck squamous cell carcinoma. ESMO Open. 2021 Apr;6(2):100075. doi: 10.1016/j.esmoop.2021.100075. Epub 2021 Mar 10. PMID 33714009